CLINICAL TRIAL: NCT01967069
Title: A Comparison of DFD01 Spray Versus Vehicle Spray in Subjects With Moderate Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1206
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFD01 Spray (Active Comparator): DFD01 Spray twice daily
  Interventions: Drug: DFD01 Spray
- Vehicle Spray (Placebo Comparator): Vehicle Spray twice daily
  Interventions: Drug: Vehicle Spray

INTERVENTIONS:
Drug: DFD01 Spray
  Arms: DFD01 Spray
Drug: Vehicle Spray
  Arms: Vehicle Spray

SUMMARY:
The objectives of this study are to compare the efficacy and safety of DFD01 Spray to Vehicle Spray for topical treatment of moderate plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

Subjects must present with a clinical diagnosis of stable (at least 3 months) plaque-type psoriasis.

Subjects with psoriasis involving 10 to 20% BSA, not including the face, scalp, groin, axillae and other intertriginous areas.

Subjects must have an IGA grade of 3 (moderate) at the Baseline Visit

Exclusion Criteria:

Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis Other inflammatory skin disease that may confound the evaluation of the plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis).

Presence of pigmentation, extensive scarring, or pigmented lesions or sunburn which could interfere with the rating of efficacy parameters.

History of psoriasis unresponsive to topical treatments. History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.

Use within 180 days prior to Baseline Visit of biologic treatment for psoriasis (e.g., infliximab, adalimumab, etanercept, ustekinumab, or alefacept).

Have received treatment for any type of cancer within 5 years of the Baseline Visit except skin cancer and cervical cancer (in situ) are allowed within 1 year of the Baseline Visit.

Use within 60 days prior to the Baseline Visit of: 1) immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), 2) systemic antipsoriatic treatment (e.g., methotrexate, cyclosporine, hydroxyurea) or 3) oral retinoids (e.g., acitretin, isotretinoin).

Use within 30 days prior to the Baseline Visit of: 1) systemic steroids, 2) PUVA therapy, 3) systemic anti-inflammatory agents (e.g., mycophenolate mofetil, sulfasalazine, 6-thioguanine), or 4) UVB therapy. Inhaled, intraocular, and intranasal steroids are allowed.

Use within 14 days prior to the Baseline Visit of: 1) topical antipsoriatic drugs (e.g., salicylic acid, anthralin, coal tar, calcipotriene), 2) topical retinoids (e.g., tazarotene, tretinoin) or 3) topical corticosteroids.

Require use of beta blockers, lithium, ACE inhibitors, and/or NSAIDs (indomethacin, ibuprofen, aspirin, naproxen) with a medical history that these medications affect the subject's psoriasis, except if the subject has been using the medication routinely during the 180 days prior to the Baseline Visit, these medications are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Hudson Dermatology/Clinical Research Advantage, Tempe, Arizona
  - Dermatology Specialists, Inc., Oceanside, California
  - University Clinical Trials, Inc, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Skin Care Research, Inc., Boca Raton, Florida
  - MOORE Clinical Research, Inc., Brandon, Florida
  - FXM Research Corop., Miami, Florida
  - Dr. Tory P. Sullivan, MD, PA, North Miami Beach, Florida
  - Augusta Centre for Dermatology and Skin Renewal, LLC, Augusta, Georgia
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - MLFKnuckles, MD, PSC, Corbin, Kentucky
  - Shondra L. Smith, MD Dermatology & Advanced Aesthetics, Lake Charles, Louisiana
  - Henry Ford Medical Center, New Center One, Detroit, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Skin Specialists P.C., Omaha, Nebraska
  - Bettencourt Skin Center, Henderson, Nevada
  - Skin Search of Rochester, Inc., Rochester, New York
  - Radiant Research, Inc., Cincinnati, Ohio
  - Brodell Medical, Inc., Warren, Ohio
  - Paddington Testing Company, Inc., Philadelphia, Pennsylvania
  - Center for Clinical Studies, LTD, LLP, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Progressive Clinical Reesearch, PA, San Antonio, Texas
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Eastern Washington Dermatology, Walla Walla, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- DFD01 Spray: DFD01 Spray twice daily
  DFD01 Spray
- Vehicle Spray: Vehicle Spray twice daily
  Vehicle Spray
Period: Overall Study
Arm/Group | DFD01 Spray | Vehicle Spray
Started | 182 | 95
Completed | 174 | 87
Not Completed | 8 | 8
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD01 Spray | Vehicle Spray | Total
Number analyzed (Participants) | 182 | 95 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (14.72) | 49.9 (12.90) | 50.2 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 37 | 105
  Male | 114 | 58 | 172
Region of Enrollment [Number; unit: participants]
  United States | 182 | 95 | 277
% Body Surface Area [Mean (Standard Deviation); unit: Percent] | 13.7 (3.72) | 13.4 (3.49) | 13.6 (3.64)
Participants with Moderate Psoriasis According to the Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] | 182 | 95 | 277

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success According to the Investigator's Global Assessment (IGA)
Description: IGA of clear or almost clear
Time Frame: Day 15
Population: Intent to Treat
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | DFD01 Spray | Vehicle Spray
Number analyzed (Participants) | 182 | 95
percentage of subjects | 21.50 [15.5 to 27.5] | 7.4 [2.1 to 12.7]

ADVERSE EVENTS:
Description: Three subjects in the betamethasone dipropionate spray 0.05% group and two subjects in the vehicle spray group had no post-baseline safety evaluations.
Arm/Group | DFD01 Spray | Vehicle Spray
Serious Adverse Events (participants affected / at risk) | 1/179 | 2/93
Other Adverse Events (participants affected / at risk) | 17/179 | 24/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD01 Spray (N=179) | Vehicle Spray (N=93)
Upper Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection Right Foot (Infections and infestations) | 0 (0) | 1 (1)
Exacerbation of Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD01 Spray (N=179) | Vehicle Spray (N=93)
Application Site Pain (General disorders) | 5 (5) | 10 (10)
Application Site Pruritus (General disorders) | 12 (12) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days